CLINICAL TRIAL: NCT05238740
Title: Comparison of Radiographic Fusion Rate and Clinical Outcome of Anterior Lumbar and Extreme Lateral Interbody Fusion Performed With Either Recombinant Human Bone Morphogenetic Protein-2 or ViviGen® Cellular Bone Matrix, a Prospective Randomised Assessor Blind, Monocentric Trial
Brief Title: Comparison of Radiographic Fusion Rate and Clinical Outcome of ALIF and XLIF Performed With Either Recombinant Human Bone Morphogenetic Protein-2 or ViviGen®
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenhofgruppe AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021-02219
Record Dates: First submitted 2022-01-07; First posted 2022-02-14 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Spondylosis; Spondylolisthesis; Degenerative Disc Disease
Keywords: ViviGen; Radiographic fusion rate; Anterior lumbar interbody fusion; Recombinant human bone morphogenetic protein-2; Spondylosis; Spondylolisthesis; Degenerative Disc Disease; Extreme lateral interbody fusion
MeSH Terms: conditions — Spondylosis; Spondylolisthesis; Intervertebral Disc Degeneration | interventions — Bone Morphogenetic Protein 2

STUDY DESIGN:
Intervention Model Description: The study is a prospective randomized assessor blind monocentric trial. It aims for non-inferiority.
Who Masked: Outcomes Assessor
Masking Description: The CT Reviewer and data analysts, will be blinded as to which bone graft treatment the patient received. Blinding is ensured by coding the electronic case report forms (eCRFs)/ database and images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group 5-5.4 cc ViviGen® (Active Comparator): Biological: 5-5.4 cc ViviGen® The ALIF or XLIF fusion patients assigned to this group will receive 5-5.4 cc ViviGen®
  Interventions: Other: ViviGen®
- Control group 4-6mg rhBMP-2 (Active Comparator): Biological: 4-6mg rhBMP-2 The ALIF or XLIF fusion patients assigned to this group will receive 4-6mg rhBMP-2
  Interventions: Other: rhBMP-2

INTERVENTIONS:
Other: ViviGen® — It will investigate the radiological and clinical outcome of ALIF procedure L5/S1 and XLIF L4/L5 procedure using two arms/ treatments, namely either ViviGen® Bone Matrix (intervention group) or rhBMP-2 (control group). ViviGen®/ rhBMP-2 ratio will be 1:1.
  Arms: Intervention group 5-5.4 cc ViviGen®
Other: rhBMP-2 — It will investigate the radiological and clinical outcome of ALIF procedure L5/S1 and XLIF L4/L5 procedure using two arms/ treatments, namely either ViviGen® Bone Matrix (intervention group) or rhBMP-2 (control group). ViviGen®/ rhBMP-2 ratio will be 1:1.
  Other Names: InductOS
  Arms: Control group 4-6mg rhBMP-2

SUMMARY:
The aim of this study is to prospectively investigate the potential for bony fusion of ViviGen® bone graft substitute in comparison to rhBMP-2 in monosegmental ALIF procedure L5/S1 and in monosegmental XLIF procedure L4/5

DETAILED DESCRIPTION:
The investigator hypothesize that

- The bony fusion rate on a 12-month CT scan (or earlier at 6-month CT scan) is less than 10% lower in the intervention group compared to the bony fusion rate in the control group

For patients included in the study, all follow-up is recorded, with regards to radiological and clinical outcome. Follow up will be evaluated after 14 days, 6 weeks, 6 and 12 months. Last follow up will be 1 year after surgery.

ELIGIBILITY:
Inclusion criteria:

Patients who have an indication for a monosegmental ALIF procedure on the L5/S1 segment or a monosegmental XLIF procedure on L4/5 (both ALIF and XLIF procedure with or without an additional pedicular stabilisation), e.g., treating conditions such as spondylosis, spondylolisthesis and degenerative disc disorders with back and/or leg pain

* Patients must be 18 - 70 years of age
* Patients must have understood and signed the study information and the informed consent form
* Patients are willing and able to complete scheduled follow-up evaluations / questionnaires as described in the Informed Consent

Exclusion criteria:

* Patients under 18 years and over 70 years of age
* Patients with tumour / spine trauma / known bone disease / Parkinson's disease and similar CNS disorders / diseases or injuries of the peripheral nerves
* Other procedures or segment than mentioned in the inclusion citeriaAdditional planed spine surgeries after index surgery
* Current smoking
* Pregnant or breastfeeding patients (or patient planning a pregnancy within one year after surgery)
* Insufficient language skills in German
* Inability to give informed consent
* Refusal to participate in the study, unsigned study consent
* Participation in another interventional study within the 30 days preceding and during the present study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of interbody bony fusion in the treated patients confirmed at 12-month CT or earlier at 6-month CT using Brantigan, Steffee, Fraser (BSF) | 6 or 12 months after intervention
  The rate of interbody bony fusion will be assessed by computed tomography and then by a radiologist 6 or 12 months after the intervention.
  Modified Brantigan, Steffee, Fraser (BSF) classification of interbody fusion success will be defined as follows:
  BSF-1: Radiographical pseudarthrosis is indicated by collapse of the construct, loss of disc height, vertebral slip, broken screws, displacement of the Synfix cage, or significant resorption of the bone graft, or lucency visible around the periphery of the graft or cage.
  BSF-2: Radiographical locked pseudarthrosis is indicated by lucency visible in the middle of the cages with solid bone growing into the cage from each vertebral endplate.
  BSF-3: Radiographical fusion: bone bridges at least half of the fusion area with at least the density originally achieved at surgery. Radiographical fusion through one cage (half of the fusion area) is considered to be mechanically solid fusion even if there is lucency on the opposite side.

SECONDARY OUTCOMES:
Back pain visual analogue scale | before intervention and at 6 weeks, 6 months and 12 months after intervention
  The back pain visual analogue scale (VAS 1-10) will be assessed before intervention and at 6 weeks, 6 months and 12 months after intervention.
Leg pain visual analogue scale | before intervention and at 6 weeks, 6 months and 12 months after intervention
  The leg pain visual analogue scale (VAS 1-10) will be assessed before intervention and at 6 weeks, 6 months and 12 months after intervention.
Quality of life using a simplified Spine Tango questionnaire and the Core Outcome Measures Index (COMI Score) | before intervention and at 6 weeks, 6 months and 12 months after intervention
  Quality of life will be assessed by using a simplified Spine Tango questionnaire and the Core Outcome Measures Index (COMI Score) before intervention and at 6 weeks, 6 months and 12 months after intervention.
Disability/ limitations in the activities of daily living using a simplified Spine Tango questionnaire and the Core Outcome Measures Index (COMI Score) | before intervention and at 6 weeks, 6 months and 12 months after intervention
  Disability / limitations in the activities of daily living will be assessed by using a simplified Spine Tango questionnaire and the Core Outcome Measures Index (COMI Score) before intervention and at 6 weeks, 6 months and 12 months after intervention.
Disability/ limitations at the workplace using a simplified Spine Tango questionnaire and the Core Outcome Measures Index (COMI Score) | before intervention and at 6 weeks, 6 months and 12 months after intervention
  Disability / limitations at the workplace will be assessed by using a simplified Spine Tango questionnaire and the Core Outcome Measures Index (COMI Score) before intervention and at 6 weeks, 6 months and 12 months after intervention.
Patient satisfaction using a simplified Spine Tango questionnaire and the Core Outcome Measures Index (COMI Score) | 6 weeks, 6 months and 12 months after intervention
  Patient satisfaction will be assessed by using a simplified Spine Tango questionnaire and the Core Outcome Measures Index (COMI Score) at 6 weeks, 6 months and 12 months after intervention.
Complication / side effects using a simplified Spine Tango questionnaire and the Core Outcome Measures Index (COMI Score) | 14 days, 6 weeks, 6 months and 12 months after intervention
  Complication / side effects will be assessed by using a simplified Spine Tango questionnaire and the Core Outcome Measures Index (COMI Score) at 14 days, 6 weeks, 6 months and 12 months after intervention.

OTHER OUTCOMES:
Healthcare-costs using hospitalisation length of stay (LOS), occurrence and therapy of side effects/ adverse events and necessary revision operations | 12 months after intervention
  Healthcare-costs will be assessed by using hospitalisation length of stay (LOS), occurrence and therapy of side effects/ adverse events and necessary revision operations at 12 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Diel Peter, Dr. med., Principal Investigator — Orthopädie Sonnenhof, Bern
Locations (1):
- Orthopädie Sonnenhof, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arrington ED, Smith WJ, Chambers HG, Bucknell AL, Davino NA. Complications of iliac crest bone graft harvesting. Clin Orthop Relat Res. 1996 Aug;(329):300-9. doi: 10.1097/00003086-199608000-00037. PMID 8769465
- [Background] Birmingham E, Niebur GL, McHugh PE, Shaw G, Barry FP, McNamara LM. Osteogenic differentiation of mesenchymal stem cells is regulated by osteocyte and osteoblast cells in a simplified bone niche. Eur Cell Mater. 2012 Jan 12;23:13-27. doi: 10.22203/ecm.v023a02. PMID 22241610
- [Background] Johnstone B, Zhang N, Waldorff EI, Semler E, Dasgupta A, Betsch M, Punsalan P, Cho H, Ryaby JT, Yoo J. A Comparative Evaluation of Commercially Available Cell-Based Allografts in a Rat Spinal Fusion Model. Int J Spine Surg. 2020 Apr 30;14(2):213-221. doi: 10.14444/7026. eCollection 2020 Apr. PMID 32355628
- [Background] Kadam A, Millhouse PW, Kepler CK, Radcliff KE, Fehlings MG, Janssen ME, Sasso RC, Benedict JJ, Vaccaro AR. Bone substitutes and expanders in Spine Surgery: A review of their fusion efficacies. Int J Spine Surg. 2016 Sep 22;10:33. doi: 10.14444/3033. eCollection 2016. PMID 27909654
- [Background] Manzur M, Virk SS, Jivanelli B, Vaishnav AS, McAnany SJ, Albert TJ, Iyer S, Gang CH, Qureshi S. The rate of fusion for stand-alone anterior lumbar interbody fusion: a systematic review. Spine J. 2019 Jul;19(7):1294-1301. doi: 10.1016/j.spinee.2019.03.001. Epub 2019 Mar 11. PMID 30872148
- [Background] Singh K, Ahmadinia K, Park DK, Nandyala SV, Marquez-Lara A, Patel AA, Fineberg SJ. Complications of spinal fusion with utilization of bone morphogenetic protein: a systematic review of the literature. Spine (Phila Pa 1976). 2014 Jan 1;39(1):91-101. doi: 10.1097/BRS.0000000000000004. PMID 24026158
- [Background] Wetzell B, McLean JB, Moore MA, Kondragunta V, Dorsch K. A large database study of hospitalization charges and follow-up re-admissions in US lumbar fusion surgeries using a cellular bone allograft (CBA) versus recombinant human bone morphogenetic protein-2 (rhBMP-2). J Orthop Surg Res. 2020 Nov 19;15(1):544. doi: 10.1186/s13018-020-02078-7. PMID 33213484